CLINICAL TRIAL: NCT05215587
Title: Scandinavian Trial of Uncomplicated Aortic Dissection Therapy
Acronym: SUNDAY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Swedish Research Council (Other Government); Swedish Heart Lung Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8240
Record Dates: First submitted 2022-01-17; First posted 2022-01-31 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-03

CONDITIONS: Aortic Dissection
Keywords: Aortic; dissection; TEVAR; endovascular; vascular
MeSH Terms: conditions — Aortic Dissection | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Intervention Model Description: The trial is a randomized, open label, clinical trial with parallel assignment of patients in multiple centres in Denmark, Sweden, Norway, Finland, Iceland, New Zealand, and the Netherlands. Recruited subjects will undergo stratified randomization based on the centre to either a control or intervention arm.
Who Masked: Outcomes Assessor
Masking Description: Data are collected and stored using the Research Electronic Data Capture (REDCap) software. Overall access is granted only to the Data and Safety Monitoring Committee and the Trial Steering Committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Medical Therapy (No Intervention): Patients will be treated with standard medical therapy, i.e., antihypertensives, pulse-rate regulators, and pain medication.
- Stent Therapy (Active Comparator): Patients will be treated with both standard medical therapy, in addition to placement of a thoracic endovascular aortic repair stent graft.
  Interventions: Device: TEVAR

INTERVENTIONS:
Device: TEVAR — A TEVAR stent graft will be placed in the descending aorta in order to cover the primary entry of the dissection.
  Other Names: Thoracic aortic endovascular repair stent graft
  Arms: Stent Therapy

SUMMARY:
The introduction of thoracic endovascular aortic repair (TEVAR) in 1994 has radically changed the treatment of thoracic aortic pathology, and TEVAR is now the recommended therapy for "complicated" TBADs and other thoracic aorta diseases. To date, the use of TEVAR in the treatment of "uncomplicated" dissections (uTBAD) is uncertain, although it is presumed that a prophylactic procedure can prevent later complex surgery and early death. Several analyses have found that TEVAR confers improved aortic remodeling and possibly survival, although these were underpowered for this specific outcome. In addition, there are several reports regarding the uncertain benefit or harm of this intervention in the vascular surgery community. Put another way, there is equipoise, and the need for robust evidence in the form of a randomized clinical trial has been clearly iterated by the European Society of Vascular Surgery.

This randomized, open-label, two-armed controlled study directly addresses this question of whether TEVAR alters 5-year survival among patients with an uTBAD. Patients will be randomized to either standard medical therapy (SMT) alone or TEVAR in addition to SMT. The primary outcome is 5-year survival, while secondary outcomes include aortic-related mortality, neurological events, quality of life, costs, re interventions and readmissions. in addition, subgroup analyses based on the extent of treatment.

Sample size calculations based on previous reports indicate the need to include approximately 554 patients. Patients will be recruited from multiple centres in Scandinavia. Based on the population (24 million) and incidence of uTBAD (approximately 480 per year), and depending on the total number of participating centres, a conservative estimate of two to three years is required for enrolment.

DETAILED DESCRIPTION:
This randomized, open-label, two-armed controlled study addresses the question of whether thoracic endovascular aortic repair (TEVAR) alters 5-year survival among patients with an uncomplicated Stanford type-B aortic dissection (uTBAD). Patients will be randomized to either standard medical therapy (SMT) alone or TEVAR in addition to SMT. The primary outcome is 5-year survival, while secondary outcomes include aortic-related mortality, neurological events, quality of life, costs, re interventions and readmissions. in addition, subgroup analyses based on the extent of treatment.

Primary hypothesis:

The null hypothesis for this trial states that the five-year survival results for patients treated with either SMT or SMT + TEVAR are equivalent.

2. Background

The incidence of a Stanford type-B thoracic aortic dissection (TBAD) is estimated at 3.9 - 6.0 per 100,000 person years, although this may be an underestimate. These account for approximately 30-40% of all types of aorta dissection. The diagnosis of TBAD is further classified with respect to time: acute, ≤ 14 days, subacute, 15-90 days, and chronic, > 90 days. Approximately 40-50% of ABDs are considered complicated which, according to the European Society of Vascular Surgery, is defined as the presence of one or more of the following: rupture and/or hypotension/shock, organ malperfusion, rapid aortic expansion, paraplegia/paraparesis, peri-aortic haematoma, or intractable pain or hypertension. In the absence of these complications, the dissection is considered uncomplicated. In-hospital survival for these patients has been reported as approximately 90%.

The management of TBADs is dependent upon the above-mentioned factors, i.e., complicated or uncomplicated, acute or chronic, as well as accompanying comorbidities. An underlying and universal component for all these patients is optimal medical therapy, which includes antihypertensive therapy, typically beta-blockers, in order to mitigate aortic wall stress and false lumen pressures, as well as pain relief. Furthermore, lifestyle improvements and cardiovascular risk profile modification are recommended.

The introduction of thoracic endovascular aortic repair (TEVAR) in 1994 radically changed the treatment of thoracic aortic pathology, and TEVAR is now the recommended therapy for complicated TBADs, thoracic aortic aneurysms, and traumatic thoracic transections, among others. To date, the use of TEVAR in the treatment of uncomplicated TBAD is uncertain, if not controversial. Several analyses have found that TEVAR confers improved aortic remodeling and possibly survival, albeit with the implied and inherent procedural risks of intervention, including paraplegia, retrograde dissection, and death.

There are two relevant randomized clinical trials (RCTs), addressing the issue of early TEVAR among TBAD patients. The Acute Dissection: Stent graft OR Best medical therapy (ADSORB) trial, notably underpowered, randomized a total of 61 patients from 17 European centres with acute uTBAD. There were no aortic ruptures at 1-year in either arm of the trial, while TEVAR was associated with improved thrombosis of the false lumen and reduction of its lumen. The Investigation of Stent Grafts in Aortic Dissection (INSTEAD) trial included 140 patients in the subacute phase. The overall survival at two years was statistically equivalent, 95.6% in the medical arm and 88.9% in the TEVAR plus medicine group. The long-terms results from the extended INSTEAD-XL found a non-significant absolute reduction in all-cause mortality of 8.2% at five years for those patients who underwent TEVAR.

The conclusions from the retrospective and above-mentioned RCTs have not been persuasive enough for the European Society of Vascular Surgery to render a higher recommendation than "TEVAR may be selectively considered" for those patients presenting with uncomplicated type B aortic dissections. This is furthermore echoed by a recent international survey regarding preferred treatment of uTBAD, in which 54.8% of respondents answered that they do not routinely use TEVAR, as opposed to 37.4% who prefer this strategy; moreover, 88.6% of respondents agreed that equipoise was present and that an RCT was warranted.

Research Objectives

Primary Objective

• To compare the overall survival at five years between subjects treated with SMT or SMT + subacute TEVAR.

Secondary Objectives

* To compare the risk of aortic-related mortality.
* To compare the risk of neurological injury, including stroke or paraplegia.
* To compare the proportion and indication of subjects who underwent an aortic intervention within 5 years due to development of an aortic complication.
* To compare the number of disease-related readmissions during follow-up.
* To compare, based on subgroup analyses, whether extent of TEVAR is associated with either improved survival or neurological injury.
* To compare the associated risk of reinterventions, including those subjects who were initially randomized to SMT and subsequently required an aortic intervention.
* To compare the associated changes in quality-of-life.
* To compare the 10-year overall survival and aortic-related mortality.
* To compare the costs.

Endpoint Definitions

Primary endpoint:

All-cause mortality.

Secondary endpoints:

Aortic-related mortality: Death as a result from aortic rupture or organ malperfusion, or death due to aortic intervention.

Aortic intervention: Any open surgical or endovascular intervention performed in any anatomical location, performed for the following indications, which are related to the aortic pathology: aneurysmal degeneration, visceral ischemia, lower extremity ischemia, rupture, or any of the criteria listed above under the definition of a complicated TBAD.

Neurological injury: These are divided into two categories: cerebrovascular accidents (CVA) and spinal cord ischemia (SCI). CVAs are defined according to the Society for Vascular Surgery reporting standards and classified as any central neurological complication, ischemic and hemorrhagic. For this project, the modified Rankin scale will be used for classifying stroke severity. Spinal cord ischemia is defined as either ischemic or hemorrhagic resulting in paraparesis or paraplegia. The modified Tarlov scoring scale will be used for the grading of any spinal cord injuries.

Reintervention: Any open or endovascular intervention after the original TEVAR procedure that was related to the dissection. These should be categorized as either planned reintervention, e.g., a staged procedure, or unplanned, which indicates a complication from the original procedure, a failure of the device, or progression of disease.

Quality of life: The quality of life will be assessed with the three following self-assessment forms:

1. The EuroQOL-5D-5L instrument from the EuroQol Group, comprised of five dimensions with five levels of scoring that can be combined into a five-digit number of description.
2. The Hospital and Anxiety Depression Score (HADS).
3. The 12-Item Short-Form (12-SF) Health Survey.

Economic evaluation: The economic evaluation will be performed from a payer/healthcare point of view, including resource use associated with healthcare, intervention and medication, whereas broader potential consequences for society, i.e., effects on productivity, will not be included. During the course of the trial, the accumulated costs will be measured per treatment arm from the participating hospital´s administrative/controlling/billing systems. As far as possible, the following resource use items will be included and captured as accumulated costs from the hospital's cost-per- subject system on all outpatient and inpatient visits:

* costs for healthcare staff
* subject -specific costs for primary and secondary endovascular and surgical procedures postoperative care unit costs
* costs of drugs during surgery and postoperative care
* costs of anaesthetic procedures and blood transfusions
* additional diagnostic procedures from the radiology and clinical physiology departments and from clinical chemistry.

The costs for healthcare staff will comprise the full wage costs, including costs for social security. Costs for each endovascular and surgical procedure will be retrieved individually, and, as far as possible, be based on the price per minute according to the hospital's cost-per- subject systems.

Changes in health status will be assessed in terms of quality-adjusted life-years (QALYs), which combine the time spent in a specific health state with the corresponding self-assessed health-related quality of life (HRQoL), as derived from the EuroQOL EQ-5D-5L questionnaire. Time is measured in years and the HRQoL is measured on an index scale ranging from 0 (equivalent to being dead) to 1 (best possible health state). The total number of QALYs will be calculated by multiplying the HRQoL index score (QALY weight) by the time spent in each health state. Group differences in total costs will be calculated and divided by the difference in QALYs in the interval from baseline until end of study, and the incremental cost-effectiveness ratio will be calculated as follows:

(CostTEVAR -CostSMT)/(QALYsTEVAR - QALYsSMT)=ΔCost/ΔQALY.

Rationale for objectives and endpoint selection

Despite evidence from retrospective and descriptive studies suggesting long-term benefits for early TEVAR intervention among uTBAD subjects, the underlying unanswered question is whether TEVAR confers a benefit of survival. The two previous RCTs, mentioned above, were underpowered to address this issue. Despite potential theoretical and procedural advantages of various composite endpoints, it was determined that a trial based on a clearly expressed question with a binary outcome will have the most clinical impact. Similarly, focus on the albeit interesting, but not essential, endpoint of aortic morphological changes and imaging findings, would complicate the pragmatic design of this trial.

Study Design

The trial is a randomized, open label, clinical trial with parallel assignment of subjects in multiple sites in Denmark, Sweden, Norway, Iceland, and Finland. Recruited subjects will be randomized to either SMT exclusively or TEVAR + SMT.

ELIGIBILITY:
Inclusion Criteria:

All subjects, aged 18 or greater at the time of informed consent, admitted or referred to the participating vascular surgery site with an uTBAD of less than four weeks duration.

Exclusion Criteria:

* Subjects with no signed informed consent.
* Subjects presenting with a complicated type B aortic dissection according to the above definition.
* Subjects previously treated in their descending aorta, either open surgery or TEVAR.
* Subjects with pre-existing thoracoabdominal aortic aneurysm.
* Subjects with other aortic pathology with an indication for intervention that requires TEVAR.
* Subjects with traumatic aortic dissections.
* Subjects with an established connective tissue disease at the time of randomization, including but not limited to Marfans and Loeys-Dietz syndrome.
* Subjects with a clinically estimated life expectancy < 2 years.
* Subjects with dementia.
* Pregnant or nursing subjects.
* Subjects with current sepsis.
* Subjects currently participating in other clinical interventional trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | Five years
  Overall survival

SECONDARY OUTCOMES:
Aortic-related mortality | Five years
  Death as a result from aortic rupture or organ malperfusion, or death due to aortic intervention.
Neurological injury | Five years
  Cerebrovascular accidents and/or spinal cord ischemia
Reintervention | Five years
  The number of open or endovascular interventions after the original TEVAR, including crossovers, that were related to the dissection. Categorised as planned or unplanned.
EuroQOL-5D-5L | Five years
  Quality of life
Hospital Anxiety and Depression Score | Five years
  Psychological distress
12-Item Short Form Health Survey | Five years
  Physical and mental health functioning

CONTACTS AND LOCATIONS:
Overall Officials: Jacob W Budtz-Lilly, MD PhD, Principal Investigator — Aarhus University Hospital; Kevin Mani, MD PhD, Principal Investigator — Uppsala University Hospital
Locations (28):
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Copenhagen University Hospital, Rigshospital, Copenhagen
  - Odense University Hospital, Odense
- Finland (5):
  - Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- Landspitali University Hospital, Reykjavik, Iceland
- Netherlands (7):
  - Amsterdam University Medical Center (AUMC), Amsterdam
  - University Medical Center Groningen (UMCG), Groningen
  - Leiden University Medical Center (LUMC), Leiden
  - Maastricht University Medical Center (MUMC), Maastricht
  - Radboud University Medical Center (Radboudumc), Nijmegen
  - Erasmus Medical Center (EMC), Rotterdam
  - University Medical Center Utrecht (UMCU), Utrecht
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
  - University Hospital Nord, Tromsø
  - St Olavs Hospital, Trondheim
- Sweden (7):
  - Sahlgrenska University Hospital, Gothenburg
  - Linköping University Hospital, Linköping
  - Skånes University Hospital, Malmo
  - Örebro University Hospital, Örebro
  - Karolinska University Hospital, Stockholm
  - Sodersjukhuset, Stockholm
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual patient data with other researchers outside the trial.

REFERENCES:
- [Background] Rudolph C, Lindberg BR, Resch T, Mani K, Bjorkman P, Laxdal EH, Stovring H, Beck HM, Eriksson G, Budtz-Lilly J. Scandinavian trial of uncomplicated aortic dissection therapy: study protocol for a randomized controlled trial. Trials. 2023 Mar 23;24(1):217. doi: 10.1186/s13063-023-07255-7. PMID 36949478
- See also: Homepage — https://www.sundaytrial.dk